CLINICAL TRIAL: NCT02709837
Title: Impact of Food Process and Mastication on Nutrient Bioavailability
Acronym: DREAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: Centre de Recherche en Nutrition Humaine d'Auvergne (Other Government)
Responsible Party: Principal Investigator, Yves Boirie, Professor, Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: AU 1030; 2013-A00096-39 (Other: Comité de Protection des Personnes Sud-Est 6)
Record Dates: First submitted 2016-02-25; First posted 2016-03-16 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Nutrition
Keywords: bioavailability; amino acid; carnosine; lycopene; mastication; meat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Poorly cooked meat-Good chewing (Active Comparator): Meat cooked 10min at 75°C, chewing without appliance
  Interventions: Other: Nutritional
- Highly cooked meat-Good chewing (Active Comparator): Meat cooked 45min at 90°C, chewing without appliance
  Interventions: Other: Nutritional
- Poorly cooked meat-Bad chewing (Active Comparator): Meat cooked 10min at 75°C, chewing with appliance
  Interventions: Other: Nutritional
- Highly cooked meat-Bad chewing (Active Comparator): Meat cooked 45min at 90°C, chewing with appliance
  Interventions: Other: Nutritional

INTERVENTIONS:
Other: Nutritional

SUMMARY:
This project aims at assessing

* the impact of heat treatment on the bioavailability of meat carnosine and amino acids,
* the interaction between masticatory efficiency and heat treatment of meat on the bioavailability of carnosine and amino acids
* the effect of dietary calcium on tomato lycopene bioavailability.

DETAILED DESCRIPTION:
This cross-over study (double 5x5 latin square design) includes 10 young healthy subjects (5 males, 5 females).These subjects are studied in two different situations: a situation of good chewing efficiency, and a situation of disturbed chewing. This second situation is simulated by the wearing an occlusal appliance interfering with chewing and experimentally leading to poor masticatory efficiency. The overall study is conducted in two distinct protocols. The first protocol "Food bolus" is dedicated to the study of the rheological properties of the food bolus including analysis of the release of amino acids and bioactive peptides (secondary objective). The second protocol "Bioavailability" is the study of the bioavailability of bioactive compounds target (main objective). Each volunteer participates in both protocols. The sessions, with or without occlusal appliance, are randomized individually for each subject. Each subject is his own control and confounding factors related to individual variability of mastication and the general functioning of the digestive tract are therefore minimized.

Meat model was pork (Longissimus dorsi). Meat was sliced 2 cm thick, and two types of cooking were applied: 10 min cooking at 75 ° C and 45 min cooking at 90 °C. Meat was presented to volunteers in the form of pre-calibrated cubes (2x2x2 cm) of about 7 g.

Protocol 1: Sampling for "food bolus" study This part of the study allowed a complete description of the physical / rheological properties of bolus after good or poor mastication of the pork meat cooked according to the 2 previously described conditions. The analysis of these properties is followed all along the chewing sequence, until bolus swallowing. For that, boli are collected at different moments during the sequence of mastication. Subjects stopped chewing when indicated by the experimenter, and spat out the entire bolus with the saliva. This protocol also allows the release of carnosine and amino acids from the meat matrix during mastication to be studied.

Protocol 2: Sampling for 'bioavailability' study The volunteers participated in five sampling days. The determination of the kinetics of appearance in peripheral blood of targeted bioactive compounds (carnosine, lycopene) as well as the release of all amino acids, is done after ingestion of a mixed meal (meat, tomato, pasta), under conditions of normal or poor chewing. Meal is prepared from 100 g of cooked meat (low cooking or high cooking meat), 40 g of tomato puree, 10 ml of olive oil, and 80 g of raw pasta. An additional meal containing calcium is tested in normal chewing condition with low cooking meat. Meals are tested on different days. These days are spaced by at least 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women
2. Women with contraception considered reliable by the investigator
3. 20 ≤ age ≤ 30 years
4. Weight: ≥ 50kg
5. Good general health
6. Normal biological balance
7. Body mass index : 20 ≤ BMI ≤ 30
8. Good oral and dental health
9. Subjects having at least 28 teeth, tolerance for missing teeth if the number of functional units remains higher than or equal to 11, or if the number of metal rings does not exceed 4
10. Subject whose dentition makes possible a stable Class I occlusion Angle to the molar level
11. Subject considered healthy on clinical examination and medical examination
12. Person who signed the information sheet and consent
13. Person subject to a social security scheme

Exclusion Criteria:

1. HCV or HIV positive Serology
2. Biological assessment considered abnormal and not compatible with the study by the investigator.
3. Pregnant or lactating
4. medical or surgical history (judged by the investigator as not compatible with the study )
5. People with neurological problems making atypical or dysfunctional swallowing (dysphagia ...)
6. Medication may interfere with the results of the study ( muscle relaxants or psychotropic)
7. Blood donation within 8 weeks prior to the start of the study
8. Oral surgery in the previous 12 months
9. Subjects in dental care or having undergone orthodontic treatment in the previous 3 years
10. Subject suffering or having suffered in the last month of the teeth , gums or mouth in general
11. People with pain during chewing, pain in the face , mouth , jaw muscles, or loud creaking joints
12. person under guardianship or not subject to a social security scheme
13. Refusal to sign the information sheet and consent
14. Refusal to be registered with the National Volunteer File
15. Person in exclusion period another study , or who have received more than €4,500 in the year following his participation in clinical trials
16. vegetarian or vegan or person not liking meat, tomato puree or pasta 17 diet without pork 18 important alcohol ( > 2 drinks / day or 20 g alcohol / day for women and > 3 drinks / day for men ) .

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-06; Primary Completion 2013-07 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Postprandial plasma carnosine concentrations (µmole/L) | 7h
  effect of chewing efficiency and food processing
Postprandial plasma amino acid concentrations (µmol/L) | 7h
  effect of chewing efficiency and food processing
Postprandial plasma lycopene concentrations (µmol/L) | 7h
  effect of calcium addition

SECONDARY OUTCOMES:
Bolus particle size distribution (%) | <1min
  effect of chewing efficiency and food processing
Bolus hardness (N) | <1min
  effect of chewing efficiency and food processing
Bolus cohesiveness (dimensionless) | <1min
  effect of chewing efficiency and food processing
Bolus elasticity (dimensionless) | <1min
  effect of chewing efficiency and food processing
Bolus stickiness (N.s) | <1min
  effect of chewing efficiency and food processing
Bolus shear resistance (N/mm) | <1min
  effect of chewing efficiency and food processing
Carnosine concentration in food bolus (µmole/L) | <1min
  effect of chewing efficiency and food processing
Amino acid concentration in food bolus (µmol/L) | <1min
  effect of chewing efficiency and food processing